CLINICAL TRIAL: NCT06583668
Title: The Effect of Therapeutic Story on Pain, Fear and Anxiety Levels in Children With Burn Dressing
Brief Title: The Effect of Therapeutic Story on Pain, Fear and Anxiety Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Niran Coban, Asst.Prof.Dr., Okan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NSS0
Record Dates: First submitted 2024-08-27; First posted 2024-09-04 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pain; Burns; Fear; Anxiety
Keywords: Anxiety; Burn; Child; Pain; Fear
MeSH Terms: conditions — Pain; Burns; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Therapeutic Story group (Experimental): I. Assessment:Before the burn dressing II. Assessment: During burn dressing II. Assessment: After burn dressing
  Interventions: Other: Therapeutic Story
- Standard care (No Intervention): I. Assessment:Before the burn dressing II. Assessment: During burn dressing II. Assessment: After burn dressing

INTERVENTIONS:
Other: Therapeutic Story — Listening and watching the therapeutic story in digital media
  Arms: Experimental: Therapeutic Story group

SUMMARY:
Aim: The aim of this study was to evaluate the effect of therapeutic story on pain, anxiety, fear and physiological parameters in children undergoing burn dressing.

Methods: A randomised controlled trial was conducted between April 2023 and June 2024 with 60 patients who were admitted to the burn unit of a hospital in Istanbul and met the inclusion criteria. Patients in the story group (n=30) were listened to the digitised story during burn dressing, while patients in the control group (n=30) did not receive any intervention other than routine care. Data were collected using the Descriptive Characteristics Form, Child Anxiety Scale-Situation Scale, Child Fear Scale, Wong-Barker Pain Scale, Parental Satisfaction Scale (VAS) and Physiological Parameters Form.

ELIGIBILITY:
Inclusion Criteria:

* - To be between 3-6 years old,
* Consideration of the first dressing of the child in the burn centre
* 2nd degree superficial and deep burns (2nd degree burns requiring hospital treatment and high pain level)
* Percentage of burns below 10 per cent (light sedation for children with burn injuries above 10 per cent)
* Not having any chronic disease other than burns
* The child's willingness to participate in the research
* It is the absence of mental, communication problems and visual impairment.

Exclusion Criteria:

* • The child's dressing has been done in a burn center before

  * Presence of 1st and 3rd degree burn areas
  * Burn percentage is over 10%

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
The effect of therapeutic history on pain | 15 month
  Wong Barker Pain Scale The Facial Expressions Rating Scale (Wong Baker) consists of six facial expressions. The facial expressions are graded as 'No pain=0 points' and 'Unbearable pain=10 points'. It is a scale based on the child's self-report and is suitable for use in children aged 3-18 years. In this scale, pain scores are given according to the numerical values given to the faces. The lowest score is '1' and the highest score is '5'. As the score obtained from the scale increases, pain tolerance decreases and as the score decreases, tolerance increases.
  This scale was used before, during and after the burn dressing.
The effect of therapeutic history on fear | 15 month
  The scale is used to assess fear in children aged 4-10 years. The scale consists of five drawn facial expressions ranging from neutral expression (0=no anxiety) to frightened face (4=severe anxiety).
  This scale was used before, during and after the burn dressing.
The effect of therapeutic history anxiety | 15 month
  Child Anxiety Scale-Dispositional (CAS-D) Scale The Child Anxiety Scale-Dispositional (CAS-D) Scale aims to determine the anxiety levels of children aged 4-10 years. The CAS-D is shaped like a thermometer with a light bulb at the bottom and horizontal lines with intervals going upwards. In order to measure the state anxiety level, the child is asked to mark how he/she feels 'at the moment'. A transparent metre is placed over the child's rating on which ½ point increments are marked, then the ½ point increment is rounded up to the nearest number. The score can range from 0 to 10.It is determined that as the score value increases, the anxiety level increases, and as the score value decreases, the anxiety level decreases.
  This scale was used before, during and after the burn dressing.

SECONDARY OUTCOMES:
The effect of the therapeutic story applied to children on parents' anxiety levels | 15 month
  State-Trait Anxiety Scale (STAI) The scale has 20 items and is graded between 1-4. The total score obtained from the scale is between 20-80. If the score obtained from the scales is low, it indicates that the anxiety of the individual is low, and if it is high, it indicates that the anxiety of the individual is high.
The effect of therapeutic history on blood pressure/systolic -diastolic | 15 month
  Physiological Parameters Form Blood pressureof the patients were obtained with a form prepared by the investigator. Blood pressure; includes systolic and diastolic blood pressure valuesThis form was used before, during and after the burn dressing.
The effect of therapeutic history on pulse rate | 15 month
  Physiological Parameters Form pulse rate of the patients were obtained with a form prepared by the investigator. This form was used before, during and after the burn dressing.
The effect of therapeutic history on saturation levels | 15 month
  Physiological Parameters Form saturation levels of the patients were obtained with a form prepared by the investigator. This form was used before, during and after the burn dressing.

CONTACTS AND LOCATIONS:
Overall Officials: Niran ÇOBAN, Dr, Study Director — Okan University; Niran ÇOBAN, Dr, Study Director — https://www.okan.edu.tr/
Locations (1):
- Istanbul- City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Farzan R, Parvizi A, Haddadi S, Sadeh Tabarian M, Jamshidbeigi A, Samidoust P, Ghorbani Vajargah P, Mollaei A, Takasi P, Karkhah S, Firooz M, Hosseini SJ. Effects of non-pharmacological interventions on pain intensity of children with burns: A systematic review and meta-analysis. Int Wound J. 2023 Sep;20(7):2898-2913. doi: 10.1111/iwj.14134. Epub 2023 Mar 1. PMID 36859758
- [Background] Chester SJ, Stockton K, De Young A, Kipping B, Tyack Z, Griffin B, Chester RL, Kimble RM. Effectiveness of medical hypnosis for pain reduction and faster wound healing in pediatric acute burn injury: study protocol for a randomized controlled trial. Trials. 2016 Apr 29;17(1):223. doi: 10.1186/s13063-016-1346-9. PMID 27129580
- [Background] Jeffs D, Dorman D, Brown S, Files A, Graves T, Kirk E, Meredith-Neve S, Sanders J, White B, Swearingen CJ. Effect of virtual reality on adolescent pain during burn wound care. J Burn Care Res. 2014 Sep-Oct;35(5):395-408. doi: 10.1097/BCR.0000000000000019. PMID 24823326